CLINICAL TRIAL: NCT07350044
Title: A Prospective Randomized Controlled Trial Comparing Femoral Nerve Block and Combined Pericapsular Nerve Group (PENG) Plus Femoral Nerve Block for Perioperative Analgesia in Geriatric Hip Fracture Surgery
Brief Title: Comparison of Femoral Nerve Block and Combined PENG Plus Femoral Nerve Block in Geriatric Hip Surgery
Acronym: PENG-FEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, semih başkan, Doç. Prof. Dr., Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TABED1-25-1703
Record Dates: First submitted 2026-01-05; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: PENG Block; Hip Fracture Surgeries
Keywords: PENG block; Femoral block; Hip Fracture Surgeries; Pain; Opioid
MeSH Terms: conditions — Pain | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in parallel to one of two groups. One group will receive a preoperative femoral nerve block, while the other group will receive a combination of preoperative pericapsular nerve group (PENG) block and femoral nerve block. All interventions will be performed before surgery, and participants will be followed for 24 hours postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral Nerve Block (Experimental): Participants will receive a preoperative ultrasound-guided femoral nerve block performed approximately 30 minutes before surgery.
  Interventions: Procedure: Femoral Nerve Block
- PENG Block + Femoral Nerve Block (Experimental): Participants will receive a combination of preoperative ultrasound-guided pericapsular nerve group (PENG) block and femoral nerve block performed approximately 30 minutes before surgery.
  Interventions: Procedure: Pericapsular nerve group (PENG) block plus femoral nerve block

INTERVENTIONS:
Procedure: Pericapsular nerve group (PENG) block plus femoral nerve block — Combination of ultrasound-guided pericapsular nerve group (PENG) block and femoral nerve block performed preoperatively approximately 30 minutes before surgery using 20 mL of 0.25% bupivacaine for each block for perioperative analgesia.
  Arms: PENG Block + Femoral Nerve Block
Procedure: Femoral Nerve Block — Ultrasound-guided femoral nerve block performed preoperatively approximately 30 minutes before surgery using 20 mL of 0.25% bupivacaine for perioperative analgesia.
  Arms: Femoral Nerve Block

SUMMARY:
Hip fracture surgery in geriatric patients is frequently associated with severe perioperative pain, which may complicate positioning for spinal anesthesia and increase perioperative opioid requirements. Regional analgesic techniques are commonly used to improve patient comfort and reduce opioid consumption in this vulnerable population. The femoral nerve block is a well-established method for analgesia in hip surgery, while the pericapsular nerve group (PENG) block has emerged as a novel technique targeting articular branches of the hip joint with potential advantages in pain control.

This prospective randomized controlled trial aims to compare the analgesic efficacy of femoral nerve block alone versus a combined pericapsular nerve group (PENG) plus femoral nerve block in geriatric patients undergoing hip fracture surgery under spinal anesthesia. The primary outcomes include perioperative pain intensity, opioid consumption within the first 24 hours postoperatively, and the need for additional analgesia during positioning for spinal anesthesia. Secondary outcomes include spinal anesthesia procedure duration, time to sensory block onset, time to first postoperative opioid requirement, and perioperative hemodynamic parameters.

The results of this study are expected to clarify whether the addition of the PENG block to femoral nerve block provides superior perioperative analgesia and improved patient comfort compared with femoral nerve block alone in geriatric hip fracture surgery.

DETAILED DESCRIPTION:
Hip fractures represent one of the most common orthopedic emergencies in the geriatric population and are associated with significant pain, morbidity, and mortality. Effective perioperative analgesia is essential in this fragile patient group, as inadequate pain control may contribute to delayed mobilization, increased cardiopulmonary complications, delirium, and prolonged hospital stay. Traditional opioid-based analgesic strategies are frequently associated with adverse effects such as nausea, vomiting, respiratory depression, and cognitive impairment, particularly in elderly patients. Therefore, regional anesthesia techniques have gained increasing importance in hip fracture surgery.

The hip joint has a complex sensory innervation primarily derived from the femoral, obturator, and accessory obturator nerves. The femoral nerve block is a well-established technique that provides effective analgesia for hip surgery; however, it may be associated with quadriceps muscle weakness due to motor fiber involvement, potentially delaying early mobilization. The pericapsular nerve group (PENG) block, first described in 2018, selectively targets the articular branches of the femoral, obturator, and accessory obturator nerves while largely preserving motor function. Emerging evidence suggests that the PENG block may provide effective analgesia with minimal impact on quadriceps strength.

Despite these findings, the additional analgesic benefit of combining the PENG block with the femoral nerve block remains unclear. This study is designed to evaluate whether the addition of the PENG block to a standard femoral nerve block improves perioperative analgesic outcomes in elderly patients undergoing hip surgery under spinal anesthesia.

This prospective, single-center, randomized controlled trial will be conducted at Ankara Bilkent City Hospital. A total of 68 patients aged 65 years or older, classified as American Society of Anesthesiologists (ASA) physical status I-III, and scheduled for hip surgery under spinal anesthesia will be enrolled after obtaining written informed consent. Patients will be randomly allocated into two groups: Group 1 will receive a preoperative femoral nerve block, and Group 2 will receive a combination of preoperative PENG block and femoral nerve block.

All nerve blocks will be performed approximately 30 minutes before surgery in the designated block area under standard monitoring, including electrocardiography, non-invasive blood pressure measurement, and pulse oximetry. Supplemental oxygen will be administered via nasal cannula at 2 L/min. The PENG block will be performed under ultrasound guidance using an 80-mm block needle, with 20 mL of 0.25% bupivacaine injected incrementally beneath the psoas tendon between the anterior inferior iliac spine and the iliopubic eminence. The femoral nerve block will be performed under ultrasound guidance using a 50-mm block needle, with 20 mL of 0.25% bupivacaine administered incrementally around the femoral nerve.

The time to onset of sensory block will be recorded. Pain intensity will be assessed using the Visual Analog Scale (VAS) at rest and during 15° leg elevation before block placement and 30 minutes after block administration. Hemodynamic parameters, including heart rate, oxygen saturation, and systolic, diastolic, and mean arterial blood pressure, will be recorded at the same time points.

Following block assessment, patients will be transferred to the operating room and positioned in the lateral decubitus position for spinal anesthesia, with the surgical side down. VAS scores will be reassessed during positioning. If a VAS score of 4 or greater is observed during positioning, intravenous fentanyl at a dose of 1 µg/kg will be administered as rescue analgesia. Spinal anesthesia will be performed in the lateral decubitus position using 10 mg (2 mL) of hyperbaric bupivacaine. After intrathecal injection, patients will remain in the lateral position for five minutes before being positioned for surgery.

The duration of the spinal anesthesia procedure will be recorded, including patient positioning, skin antisepsis, sterile draping, intrathecal injection, and needle removal. This approach is intended to evaluate the effect of the applied peripheral nerve blocks on patient comfort and ease of positioning for spinal anesthesia.

Intraoperatively, all patients will be continuously monitored for heart rate, oxygen saturation, electrocardiography, and non-invasive (or invasive if clinically indicated) arterial blood pressure. Postoperatively, patients will be followed in the post-anesthesia care unit for 24 hours.

Postoperative pain will be assessed using VAS at 0, 2, 8, 16, and 24 hours. The time to first analgesic request, total opioid consumption within the first 24 hours, and hemodynamic parameters will be recorded. Postoperative analgesia will be standardized for all patients: intravenous paracetamol 1 g every 6 hours (maximum 4 g/day, or 3 g/day in elderly patients or those with hepatic impairment). If VAS exceeds 4 despite paracetamol administration, intravenous tramadol 50 mg will be administered as rescue analgesia, with a maximum daily dose of 300 mg. Patients will be closely monitored for opioid-related adverse effects, including sedation, nausea, vomiting, and cardiorespiratory complications.

The primary outcome of the study is the comparison of postoperative analgesic efficacy between the femoral nerve block alone and the combined PENG plus femoral nerve block, as assessed by VAS scores and opioid consumption during the first 24 hours. Secondary outcomes include intraoperative and postoperative hemodynamic stability, time to sensory block onset, ease and duration of spinal anesthesia performance, patient comfort during positioning, and time to first postoperative analgesic requirement.

The results of this study are expected to provide valuable evidence regarding the optimal regional anesthesia strategy for perioperative pain management in geriatric hip surgery patients and to contribute to improved analgesic protocols with reduced opioid exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older,
* Patients scheduled for surgery due to hip fracture,
* American Society of Anesthesiologists (ASA) physical status I-III,
* Body mass index between 18 and 40 kg/m²,
* Preoperative fasting duration of approximately 8 hours,
* Planned spinal anesthesia,
* Ability to provide written informed consent.

Exclusion Criteria:

* Age below 65 years,
* Refusal to participate in the study,
* Severe cognitive impairment, dementia, or Alzheimer's disease,
* ASA physical status IV or higher,
* Body mass index > 40 kg/m²,
* Failed spinal anesthesia or conversion to general anesthesia,
* Revision hip surgery,
* Multiple trauma patients,
* Old hip fractures (>3 weeks),
* Active malignancy receiving chemotherapy or radiotherapy,
* Active infection requiring antibiotic treatment (except prophylaxis),
* Contraindications to regional anesthesia techniques,
* Chronic steroid or immunosuppressive therapy,
* Use of anti-inflammatory drugs,
* Non-fasted patients,
* Allergy or intolerance to local anesthetics, paracetamol, tramadol, or other opioids.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score During Positioning for Spinal Anesthesia | Periprocedural: from initiation of lateral decubitus positioning for spinal anesthesia to completion of the spinal anesthetic procedure (needle withdrawal following intrathecal injection).
  To compare pain intensity during patient positioning for spinal anesthesia between the Femoral Nerve Block group and the combined Pericapsular Nerve Group (PENG) + Femoral Nerve Block group. Pain will be assessed using the Visual Analog Scale (VAS) at the time of lateral decubitus positioning for spinal anesthesia. The need for additional intravenous fentanyl during positioning will also be recorded.

SECONDARY OUTCOMES:
Postoperative Pain Scores Within the First 24 Hours | Within the first 24 hours postoperatively
  To compare postoperative pain intensity between the Femoral Nerve Block group and the combined Pericapsular Nerve Group (PENG) + Femoral Nerve Block group using the Visual Analog Scale (VAS). Pain scores will be assessed at rest and during movement at postoperative 0, 2, 8, 16, and 24 hours.
Total Opioid Consumption Within the First 24 Hours | Within the first 24 hours postoperatively.
  To compare total intravenous opioid consumption between groups within the first 24 postoperative hours. Opioid use will be recorded as cumulative tramadol consumption (mg) administered as rescue analgesia.
Hemodynamic Stability During Perioperative Period | From block application to 24 hours postoperatively
  To compare perioperative hemodynamic parameters including heart rate, systolic, diastolic, and mean arterial blood pressure, and peripheral oxygen saturation (SpO₂) between groups during the block procedure, intraoperative period, and the first 24 postoperative hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 39514540
- [Background] 38073453
- [Background] PMID: 38073453